CLINICAL TRIAL: NCT04868331
Title: Evaluation of Cardiovascular Responses in Adolescent Idiopathic Scoliosis (AIS) Girls Performing E-Fit Exercise Intervention: a Pilot Study
Brief Title: Cardiovascular Responses in Adolescent Idiopathic Scoliosis Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Rufina Lau, Senior Lecturer, Tung Wah College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-02-52-SRG190201
Record Dates: First submitted 2021-03-24; First posted 2021-04-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIS girls (Experimental): Girls between the ages of 10-16 will be recruited if they have a diagnosis of AIS.
  Interventions: Behavioral: Exercise
- Healthy Controls (Active Comparator): Healthy adolescent girls matched in age and puberty maturity without spinal deformity
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Two trials of 7-min High Intensity Interval Training (HIIT) with 12 different exercises. Each exercise lasts for 30 seconds continuously with 10 seconds rest interval.

SUMMARY:
The aims of this pilot study are to determine the metabolic demand and exercise intensity level of E-Fit exercise intervention by evaluating the cardiovascular responses in AIS girls and whether the cardiovascular responses for AIS girls performing E-Fit will behave in the same way as compared to healthy controls. We hypothesise that 1) the metabolic demand and exercise intensity of E-Fit exercise intervention is equivalent to moderate-to-vigorous level; and 2) AIS girls have different cardiovascular responses as compared to healthy controls

DETAILED DESCRIPTION:
AIS girls and age- and gender-matched healthy controls will perform the E-Fit exercise intervention for two trials and gas exchange parameters including oxygen consumption (VO2) and carbon dioxide production (VCO2) will be taken continuously during the exercise. Comparison of VO2 and VCO2 between AIS and healthy controls when performing E-Fit exercise will be made.

ELIGIBILITY:
Inclusion Criteria:

* Cobb angle greater or equal to 15 degree
* Cleared for physical activity by doctor

Exclusion Criteria:

* Cobb angle greater or equal to 40 degree, or
* Scoliosis with any known etiology, scoliosis with skeletal dysplasia, know endocrine and connective tissue abnormalities, or
* Known heart condition or other diseases that could affect the safety of exercise, or
* Eating disorders or GI malabsorption disorders, or
* Currently taking medication that affects bone or muscle metabolism

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female
Enrollment: 20 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Respiratory gas measurement | Day 1
  Breath-by-breath measurement of cardiorespiratory and gas exchange parameters to analyse oxygen consumption (VO2 in ml/min) and carbon dioxide production (VCO2 in ml/min).
Blood Pressure | Day 1
  Blood pressure (mmHg) will be measured using an electronic sphygmomanometer.
Heart rate | Day 1
  Heart rate (bpm) will be measured using a fingertip oximeter.
Oximetry | Day 1
  Peripheral capillary oxygen saturation (%) will be measured using a fingertip oximeter.

SECONDARY OUTCOMES:
Maturity assessment | Day 1
  Sexual maturity using Tanner Scale and onset of menarche will be measured.
Modified Baecke Questionnaire | Day 1
  Habitual physical activity level will be assessed by self-administered questionnaire.
Physical Activity Rating Questionnaire for Children and Youth (PARCY) | Day 1
  Physical activity level and intensity will be assessed by self-administered questionnaire.
Body height | Day 1
  Body height (cm) will be measured with standard stadiometry techniques.
Sitting height | Day 1
  Sitting height (cm) will be measured with standard stadiometry techniques.
Arm Span | Day 1
  Arm span (cm) will be measured with standard stadiometry techniques.
Body Composition | Day 1
  Percentage body fat (%), body weight (kg), lean muscle mass (kg) will be assessed using Bioelectric Impedance Analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rufina Lau, MSc, Principal Investigator — Tung Wah College
Locations (1):
- Tung Wah College, Hong Kong, Hong Kong